CLINICAL TRIAL: NCT05948774
Title: A Randomized, Double-blind, Placebo Control, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics After Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) of MT200605 for Injection in Healthy Subjects.
Brief Title: A SAD/MAD Study to Evaluate the Safety, Tolerability, PK of MT200605 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT200605-I-C01
Record Dates: First submitted 2023-06-07; First posted 2023-07-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be double-blinded for MT200605/matching placebo. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (MT200605 or placebo).Blinding will be maintained until at least the clinical phase of the study is completed. Since the outward appearance of MT200605 and Placebo is not totally same after preparations, the unblinded study nurses and Pharmacists were set up to avoid the effects of blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MT200605 for injection (Experimental): The Single Ascending Dose (SAD) and Muliple Ascending Dose (MAD) stages were built up in the study. The MT200605 in SAD and MAD following Intravenous Infusion Administration by using infusion pump in Healthy Subjects.
  Interventions: Drug: MT200605 for Injection
- MT200605 Placebo (Placebo Comparator): The Single Ascending Dose (SAD) and Muliple Ascending Dose (MAD) stages were built up in the study. The MT200605 Placebo in SAD and MAD following Intravenous Infusion Administration by using infusion pump in Healthy Subjects.
  Interventions: Drug: MT200605 Placebo

INTERVENTIONS:
Drug: MT200605 for Injection — Two stages (SAD, MAD) were designed in this study. For SAD, the MT200605 will single Intravenous (IV) infusion for 1h with the dose level as 0.15 mg/kg、0.3 mg/kg、0.6 mg/kg、0.9 mg/kg、1.2 mg/kg. For MAD, the participants will IV infusion of the MT200605 for 7 days with 2 times per day under the dose level of 0.3 mg/kg、0.6 mg/kg、1.2 mg/kg. The dosing frequency will be Q12h. The drug/placebo in day 7 will be only administrated for 1 time on morning. The infusion duration will be 1h.
  Other Names: MT200605
  Arms: MT200605 for injection
Drug: MT200605 Placebo — Two stages (SAD, MAD) were designed in this study. For SAD, the MT200605 Placebo will single Intravenous (IV) infusion for 1h with the dose level as 0.15 mg/kg、0.3 mg/kg、0.6 mg/kg、0.9 mg/kg、1.2 mg/kg. For MAD, the participants will IV infusion of the MT200605 Placebo for 7 days with 2 times per day under the dose level of 0.3 mg/kg、0.6 mg/kg、1.2 mg/kg. The dosing frequency will be Q12h. The drug/placebo in day 7 will be only administrated for 1 time on morning. The infusion duration will be 1h.
  Arms: MT200605 Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo control, Phase I clinical trial is to evaluate the Safety, Tolerability, and Pharmacokinetics after Single Ascending Dose (SAD) and multiple Ascending Dose (MAD) of MT200605 for Injection in Healthy Subjects.

The main questions it aims to answer are:

1. The safety and tolerability of MT200605 injection in health subjects
2. The Pharmacokinetic characteristic of MT200605 injction in health subjects

The study aims to recruit 60 health subjects and participants will be randomly allocate to two stages (SAD and MAD) with 36 subjects in SAD and 24 subjects in MAD stages.

The placebo will be used in this study, and the researchers will compare the placebo and test article to see if the MT200605 will be safe or well tolerated.

DETAILED DESCRIPTION:
Shaanxi Micot Technology Co. Ltd. is developing MT200605, a novel investigational synthetic small molecule tyrosine kinase B (TrkB) receptor agonist to mimic brain-derived neurotrophic factor (BDNF). It can directly bind to TrkB receptor to exert strong neuroprotective and nutritional effects and used for the indication of Treatment of brain tissue damage after cerebral ischemia-reperfusion and nerve repair after ischemic stroke.

The goal of this randomized, double-blind, placebo control, Phase I clinical trial is to evaluate the Safety, Tolerability, and Pharmacokinetics after Single Ascending Dose (SAD) and multiple Ascending Dose (MAD) of MT200605 for Injection in Healthy Subjects. The study was divided into two stages including 5 groups in SAD stage and 3 groups in MAD stage. 4 subjects were in the first corhort (C1) of SAD stage while the rest of the corhorts were 8 cases. The MT200605 and Placebo will be administrated by Intravenous injection.The dose level in SAD will be 0.15 (C1), 0.3(C2), 0.6(C3), 0.9(C4), and 1.2(C5) mg/kg. The dose level will be adjusted based on the safety and PK data of the completed SAD corhort. The dose level in MAD will be 0.3(C6), 0.6(C7), and 1.2(C8) mg/kg. The dose level will be adjusted based on the safety and PK data of the completed SAD and MAD corhort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 and ≤ 50 years of age with BMI ≥ 18.0 and ≤ 28.0 kg/m^2
2. Healthy as defined by:

   1. The absence of clinically significant illness and major surgery within 4 weeks prior to study drug administration.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Participants have no fertility plan, no sperm or egg donation plan in the next 6 months and voluntarily use effective contraception; Female subjects with negative serum pregnancy test results.
4. Can understand the study process of the clinical trial, and provide the signed ICF of joinning the clinical trial.

Exclusion Criteria:

-

Participants will be excluded from the study if any of the following applies:

1. Any clinically significant abnormal finding at physical examination.
2. Clinically significant abnormal laboratory test results or positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody at screening, or active infections.
3. Positive pregnancy test or lactating female subject.
4. Positive results of urine drug screen and breath alcohol test.
5. History of significant allergic reactions (e.g., Immediate hypersensitivity, hypersensitivity, angioedema) to any drug that the Investigator judges to be clinically significant.
6. Clinically significant ECG abnormalities (QTcF ≥ 450 ms) or vital signs abnormalities (systolic BP lower than 90 or over 140 mmHg, diastolic BP lower than 50 or over 90 mmHg, HR less than 50 or over 100 bpm) at screening.
7. History of drug abuse within 1 year prior to screening or using of the recreational drugs (such as marijuana, cocaine, phencyclidine [PCP], opioid derivatives (including Morphine, buprenorphine, methadone) or amphetamine derivatives within 3 months prior to screening.
8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 355 mL of 5% beer, or 150 mL of 12% wine, or 45 mL of 40% distilled alcohol).
9. Donation or loss of more than 500 mL blood within 2 months prior to study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months prior to screening, or plans to donate blood during the study or within 3 months after the study.
10. Estimated glomerular filtration rate (eGFR) <60 mL/min at screening (estimated with the MDRD equation).
11. Participants daily smoking of cigarettes amounts > 5 prior to the 3 months of screening, or get used to usage of nicotine-containing products, or participants who is not accept forbidden of any cigarettes products.
12. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Depot injection or implant within 3 months prior to the first dosing.
    2. Any drug or substances known to be strong inhibitors or strong inducers of CYP3A4/5, transporters of P-gp (e.g. rifampin, St, John´s Wort) within 30 days prior to the first dosing
    3. Usage of the prescription medications within 14 days prior to the first dosing.
    4. Usage of the Over-the-counter (OTC) medications (other than ≤2 g/day paracetamol [acetaminophen] or ≤ 800 mg/day ibuprofen) and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing.
13. Participants involved in the clinical trials of study drugs, marketed drug, medical devices within 90 days prior to the first dosing, or concomitant participation in an investigational study without drug or medical device administration.
14. Poor compliance or unable to comply with the relevant provisions of the research protocol, and any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-02-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events（AEs) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks.
  For SAD, AEs will be recorded and evaluated for their seriousness, severity, and relationship to the study drug.
Adverse Events（AEs) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks.
  For MAD, AEs will be recorded and evaluated for their seriousness, severity, and relationship to the study drug.
Vital signs (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks.
  Vital signs measurements including blood pressure [BP] in mmHG.
Vital signs (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks.
  Vital signs measurements including blood pressure [BP] in mmHG.
Vital signs (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including pulse rate [PR] in beats/minute.
Vital signs (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including pulse rate [PR] in beats/minute.
Vital signs (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including respiratory rate [RR] in breaths/minute.
Vital signs (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including respiratory rate [RR] in breaths/minute.
Vital signs (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including axillaty temperature [AT] in Celsius (°C).
Vital signs (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  Vital signs measurements including axillaty temperature [AT] in Celsius (°C).
12-lead electrocardiogram (ECG) recordings (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG PR Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QRS Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG RR Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QT Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QTc Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG PR Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QRS Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG RR Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QT Interval will be used to evaluate and monitor the participants.
12-lead electrocardiogram (ECG) recordings (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The ECG QTc Interval will be used to evaluate and monitor the participants.
Physical examinations-Head (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including head examination，the descriptive name of scale （inspection，palpation） will be used to report this outcome measure.
Physical examinations-Eyes (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including eyes examination，the descriptive name of scale （inspection） will be used to report this outcome measure.
Physical examinations-Ears (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including ears examination，the descriptive name of scale （auscultation） will be used to report this outcome measure.
Physical examinations-Nose (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including nose examination，the descriptive name of scale （inspection，palpation） will be used to report this outcome measure.
Physical examinations-throat (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including throat examination，the descriptive name of scale （inspection） will be used to report this outcome measure.
Physical examinations-neck (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including neck examination, the descriptive name of scale （inspection，palpation） will be used to report this outcome measure.
Physical examinations-lung (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including lung examination, the descriptive name of scale （palpation，percussion，auscultation） will be used to report this outcome measure.
Physical examinations-Abdomen (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including Abdomen examination，the descriptive name of scale （palpation） will be used to report this outcome measure.
Physical examinations-skin (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including skin examination, the descriptive name of scale （inspection，palpation） will be used to report this outcome measure.
Physical examinations-Musculoskeletal (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including musculoskeletal examination，the descriptive name of scale（inspection，palpation，percussion） will be used to report this outcome measure.
Physical examinations-Cardiovascular (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including Cardiovascular examination，the descriptive name of scale（inspection, palpation, percussion, and asking for Anamnesis）will be used to report this outcome measure.
Physical examinations-neurological (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A thorough physical examination will be performed at SAD stage, including neurological examination，the descriptive name of scale（palpation, percussion）will be used to report this outcome measure.
Physical examinations-lung (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A simple physical examination will be performed at MAD stage, including lung examination, the descriptive name of scale （palpation，percussion，auscultation） will be used to report this outcome measure.
Physical examinations-Abdomen (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A simple physical examination will be performed at MAD stage, including Abdomen examination，the descriptive name of scale （palpation） will be used to report this outcome measure.
Physical examinations-skin (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A simple physical examination will be performed at MAD stage, including skin examination, the descriptive name of scale （inspection，palpation） will be used to report this outcome measure.
Physical examinations-Cardiovascular (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  A simple physical examination will be performed at MAD stage, including Cardiovascular examination，the descriptive name of scale（inspection, palpation, percussion, and asking for Anamnesis）will be used to report this outcome measure.
Clinical laboratory test-hematology (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed, the MCH will be evaluated
Clinical laboratory test-hematology (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed,the Hematocrit will be evaluated
Clinical laboratory test-hematology (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed,the Hemoglobin will be evaluated
Clinical laboratory test-biochemistry (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The biochemistry testing will be performed, the eGFR will be evaluated
Clinical laboratory test-biochemistry (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The biochemistry testing will be performed, the serum creatinine will be evaluated
Clinical laboratory test-Urinalysis (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the urine albumin-to-creatinine ratio (UACR) will be calculated.
Clinical laboratory test-Coagulation (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the PT will be evaluated.
Clinical laboratory test-Coagulation (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the aPTT will be evaluated.
Clinical laboratory test-Coagulation (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the INR will be evaluated.
Clinical laboratory test-Cardiac Enzymes (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the TnT will be evaluated.
Clinical laboratory test-Cardiac Enzymes (SAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the TnI will be evaluated.
Clinical laboratory test-hematology (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed, the MCH will be evaluated
Clinical laboratory test-hematology (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed, the Hematocrit will be evaluated
Clinical laboratory test-hematology (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The hematology testing will be performed, the Hemoglobin will be evaluated
Clinical laboratory test-biochemistry (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The biochemistry testing will be performed, the eGFR will be evaluated
Clinical laboratory test-biochemistry (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The biochemistry testing will be performed, the serum creatinine will be evaluated
Clinical laboratory test-Urinalysis (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the urine albumin-to-creatinine ratio (UACR) will be calculated.
Clinical laboratory test-Coagulation (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the PT will be evaluated.
Clinical laboratory test-Coagulation (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the aPTT will be evaluated.
Clinical laboratory test-Coagulation (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the INR will be evaluated.
Clinical laboratory test-Cardiac Enzymes (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the TnT will be evaluated.
Clinical laboratory test-Cardiac Enzymes (MAD) | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 4 weeks
  The Urinalysis will be performed, the TnI will be evaluated.

SECONDARY OUTCOMES:
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Area under the plasma concentration versus time curve (AUC)0-t will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The AUC0-inf will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Peak Plasma Concentration (Cmax) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Time to peak drug concentration (Tmax) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Half-life (T½) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Plasma clearance (CL) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The volume of distribution (Vd) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Lambda-z (λz) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Mean Residence Time (MRT) will be calculated.
Plasma PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The AUC_%Extrap will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Cmax,ss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Tmax,ss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The AUC0-t will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The AUC0-τ will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Cmin,ss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Cav,ss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Ctrough will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The CLss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Vdss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The t1/2,ss will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Rac_AUC0-τ will be calculated.
Plasma PK of free MT200605 and total MT200605 (MAD) | Up to 2 Days.
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Rac_Cmax will be calculated.
Urine PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Ae0-t will be calculated.
Urine PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Rmax will be calculated.
Urine PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The TRmax will be calculated.
Urine PK of free MT200605 and total MT200605 (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The CLR will be calculated.
Urine PK of free MT200605 and total MT200605 (unconjugated MT200605 and total MT200605 after enzymatic hydrolysisof MT200605 glucuronide conjugate metabolits by β-glucuronidase) (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Ae0-t,ss will be calculated.
Urine PK of free MT200605 and total MT200605 (unconjugated MT200605 and total MT200605 after enzymatic hydrolysisof MT200605 glucuronide conjugate metabolits by β-glucuronidase) (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The Rmax,ss will be calculated.
Urine PK of free MT200605 and total MT200605 (unconjugated MT200605 and total MT200605 after enzymatic hydrolysisof MT200605 glucuronide conjugate metabolits by β-glucuronidase) (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The TRmax,ss will be calculated.
  CLR,ss. (The Urine of 4th Corhort in SAD will be collected and tested for Urine PK).
Urine PK of free MT200605 and total MT200605 (unconjugated MT200605 and total MT200605 after enzymatic hydrolysisof MT200605 glucuronide conjugate metabolits by β-glucuronidase) (SAD) | Up to 2 Days (the urine PK analysis only for 4th Corhort at SAD stage)
  To characterize the pharmacokinetics (PK) of MT200605 for injection in healthy adult subjects. The CLR,ss will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: RuiHua Dong, PhD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No